CLINICAL TRIAL: NCT01513720
Title: Single Dose, Two-way, Crossover, Oral Bioequivalence Study of Lamotrigine Tablets 200 mg With Lamictal® Tablets 200 mg in Healthy, Volunteers Under Fasting Condition.
Brief Title: Bioequivalence Study for Lamotrigine Tablets 200 mg Under Fasting Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AAI-US-137
Record Dates: First submitted 2012-01-17; First posted 2012-01-20 (Estimated); Last update posted 2012-01-20 (Estimated); Status verified 2002-10

CONDITIONS: Healthy
Keywords: Bioequivalence; Lamotrigine; crossover
MeSH Terms: interventions — Lamotrigine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lamotrigine Tablets 200 mg (Experimental): Lamotrigine Tablets 200 mg of Dr. Reddy's Laboratories Limited
  Interventions: Drug: Lamotrigine; Drug: Lamictal®
- Lamictal® 200 mg Tablets (Active Comparator): Lamictal® 200 mg Tablets of GlaxoSmithKline Inc
  Interventions: Drug: Lamotrigine; Drug: Lamictal®

INTERVENTIONS:
Drug: Lamotrigine — Lamotrigine Tablets 200 mg
  Other Names: Lamictal® 200 mg
Drug: Lamictal® — Lamictal® 200 mg Tablets

SUMMARY:
This is an single dose,two-way, crossover, oral bioequivalence study.

DETAILED DESCRIPTION:
The study was an single dose, two-way crossover, oral bioequivalence study of Lamotrigine tablets 200 mg of Dr. Reddy's Laboratories Limited, India comparing with that of LAMICTAL® tablets 200 mg of GlaxoSmithKline Inc, in healthy, adult, human subjects under fasting condition. 26 subjects (19 men and 7 womens) are enrolled and completed the study. The washout period is 14 days between the two periods of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females at least 18 years of age inclusive
2. Informed of the nature of the study and given written informed consent
3. Have a body weight within 15% of the appropriate range as defined in the 1983 Metropolitan Life Company tables and weighing at least 100 lbs.

Exclusion Criteria:

1. Hypersensitivity to Lamotrigine (Lamictal®) or similar compounds
2. Any history of a clinical condition which might affect drug absorption, metabolism or excretion
3. Recent history of mental illness, drug addition,drug abuse or alcoholism
4. Donation of greater than 500 ml of blood in the past 4 weeks prior to study dosing of difficulty in donating blood.
5. Received an investigational drug within the 4 weeks prior to study dosing.
6. Currently taking any prescription medication, except oral contraceptives, within the 7 days prior to study dosing or over-the -counter medication within 3 days of study dosing. This prohibition does not include vitamins or herbal preparations taken as nutritional supplements for non-therapeutics indications as judged by the attending physician.
7. Tobacco use (>5 cigarettes per day) in the 3 months prior to study dosing.
8. If female, the subjects is lactating or has a positive pregnancy test screening and prior to each of the two treatments periods. Females of child bearing potential must use a medical acceptable method of contraception throughout the entire study period and for one week after the study is completed. Medically acceptable methods or contraception that may be used by the subject and/or her partner are; oral contraceptives, progestin injection or implants, condom with spermicide, diaphragm with spermicide, IUD, vaginal spermicidal suppository, surgical sterilization of their partner(s) or abstinence. Females taking oral contraceptives must have taken them consistently for at least three months prior to receiving study medication.

Ages: 20 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2002-12; Primary Completion 2002-12 (Actual); Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
Area under curve (AUC) | Pre-dose 0.5,1,1.5,2,2.5,3,3.5,4,5,6,8,12,24,36,48,72,96,120 hours

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Ralph Scallion, MD, Principal Investigator — AAI Clinic
Locations (1):
- AAI Clinic, Quadrangle Drive, North Carolina, United States